CLINICAL TRIAL: NCT02414256
Title: PECS Block in Breast Surgery: an Observational Multicenter Study
Status: Completed | Type: Observational
Sponsor: Ospedale di Circolo - Fondazione Macchi (Other)
Responsible Party: Principal Investigator, Andrea Luigi Ambrosoli, MD, Ospedale di Circolo - Fondazione Macchi
Other Study IDs: Va-003
Record Dates: First submitted 2015-04-07; First posted 2015-04-10 (Estimated); Last update posted 2017-01-30 (Estimated); Status verified 2015-04

CONDITIONS: Postoperative Pain
Keywords: breast surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Anesthesia, Conduction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: regional anesthesia in breast surgery — In the Hospitals involved in this study are performed routinely wall blocks (PECS I-II blocks and serratus block) during breast surgery

SUMMARY:
We will enroll patients submitted to breast surgery (in and outsettings) with regional anesthesia.

The blinded observers, in the first 48 hours post-operative, will evaluate (telephone interview in outsetting) the pain intensity through the Numeric Rating Scale ( 0= no pain, 10 = worst possible pain) thereby recording the treatment procedures in accordance with usual clinical practice. At the same time we will evaluate the presence of intraoperative or postoperative complications related to regional anesthesia, the PONV rate (post-operative nausea and vomiting) and the analgesic/antiemetic therapy.

ELIGIBILITY:
Inclusion Criteria:

ASA I-II-III Patients Written Informed Consent

Exclusion Criteria:

ASA IV Active Heart Failure Coagulation Disease Chronic Pain Allergies to Local Anesthetics

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients submitted to breast surgery
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Pain Intensity Misure | 2 days

SECONDARY OUTCOMES:
Complications Regional Anesthesia Related | 1 days
PostOperative Nausea Rate | 2 days
Intraoperative Opioids Use | surgical time
Postoperative Analgesics | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Andrea L Ambrosoli, MD, Study Chair — University Hospital Varese
Locations (1):
- Department of Day Surgery Ospedale di Circolo Varese, Varese, VA, Italy